CLINICAL TRIAL: NCT04191941
Title: Adoptive Immunotherapy for Hematological Malignancy With Novel CAR-T Cells.
Brief Title: Treatment of Hematological Malignancy With Novel CAR-T Cells.
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Timmune Biotech Inc. (Industry)
Collaborators: Hunan Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-24.1
Record Dates: First submitted 2019-12-06; First posted 2019-12-10 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: B-cell Non Hodgkin Lymphoma; B-cell Acute Lymphoblastic Leukemia; Multiple Myeloma
Keywords: CD19-TriCAR-T; 1922-TriCAR-T; BCMA-TriCAR-T
MeSH Terms: conditions — Lymphoma, B-Cell; Burkitt Lymphoma; Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: Novel CAR-T Cell Therapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Novel CAR-T (Experimental): Novel CAR-T cells will be administered intravenously
  Interventions: Biological: Novel CAR-T

INTERVENTIONS:
Biological: Novel CAR-T — A conditioning chemotherapy regimen of fludarabine and cyclophosphamide may be administered, followed by a single infusion of Novel CAR-T cells

SUMMARY:
This is a single arm, open-label, early phase I study, to determine the safety and efficacy of Novel CAR-T cell therapy in Hematological Malignancy treatment.

DETAILED DESCRIPTION:
The Novel CAR-T contains either a scFv plus a PD-L1 blocker, or two scFvs, in a cytokine complex based outer memberane structure, this kind of structure enables the CAR-T cells to simultaneously target one or two targets on the tumor cell surface and enhance CAR-T cell persistence in tumor microenvironment，as well as stimulating innate T/NK cell activation and expansion.

ELIGIBILITY:
Inclusion Criteria:

1. All subjects must personally sign and date the consent form before initiating any study specific procedures or activities;
2. All subjects must be able to comply with all the scheduled procedures in the study;
3. Clear diagnosis of hematological malignancy, including B-cell Non-Hodgkin lymphoma, B-cell lymphoblastic leukemia, multiple myeloma.
4. Fufill one or more of the following criteria: Relapsed after most recent therapy; Progressive disease in standard chemotherapy; Disease progression or relapsed after ASCT;
5. At least one clear indicator for hematological malignancy monitoring;
6. Aged <70 years;
7. Expected survival ≥12 weeks;
8. Eastern cooperative oncology group (ECOG) performance status of≤3;
9. Systematic usage of immunosuppressive drug or corticosteroid must have been stopped for more than 4 weeks;
10. All other treatment induced adverse events must have been resolved to

    ≤grade 1;
11. Laboratory tests must fulfill the following criteria: ANC ≥ 1000/uL, HGB>70g/L, Platelet count ≥ 50,000/uL, Creatinine clearance ≤1.5 ULN, Serum ALT/AST ≤2.5 ULN, Total bilirubin ≤1.5 ULN (except in subjects with Gilbert's syndrome);

Exclusion Criteria:

1. Presence of fungal, bacterial, viral, or other infection that is hardly to control (defined by investigator);
2. Patients with symptomatic central nervous system metastasis, intracranial metastasis, and cancer cells found in cerebrospinal fluid are not recommended to participate in this study. Symptom free or post-treatment stable disease or disappearance of lesions should not be excluded. The specific selection is ultimately determined by the investigator;
3. Lactating women or women of childbearing age who plan to conceive during the investigational time period;
4. Active infection with hepatitis B (HBsAG positive) or hepatitis C virus (anti-HCV positive);
5. Known history of infection with HIV;
6. Subjects need systematic usage of corticosteroid;
7. Subjects need systematic usage of immunosuppressive drug;
8. Planed operation, history of other related disease, or any other related laboratory tests restrict patients for the study;
9. Other reasons the investigator consider the patient may not be suitable for the study.

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
safety (Incidence of treatment-related adverse events as assessed by CTCAE v4.03) | 3 months
  Incidence of treatment-related adverse events as assessed by CTCAE v4.03

SECONDARY OUTCOMES:
Complete response rate[CR] (Complete response rate per the revised International Working Group (IWG) Response Criteria for Malignant Lymphoma) | 3 months
  Complete response rate per the revised International Working Group (IWG) Response Criteria for Malignant Lymphoma
Partial response rate [PR] (Partial response rate per the revised International Working Group (IWG) Response Criteria) | 3 months
  Partial response rate per the revised International Working Group (IWG) Response Criteria
Duration of Response (The time from response to relapse or progression) | 24 months
  The time from response to relapse or progression
Progression Free Survival (The time from the first day of treatment to the date on which disease progresses) | 24 months
  The time from the first day of treatment to the date on which disease progresses
Overall Survival (The number of patient alive, with or without signs of cancer) | 24 months
  The number of patient alive, with or without signs of cancer

CONTACTS AND LOCATIONS:
Overall Officials: Ming Zhou, Principal Investigator — Hunan Provincial People's Hospital
Locations (1):
- Hunan Provincial People's Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No